CLINICAL TRIAL: NCT06873906
Title: Comparative Study Between Deep Parasternal Intercostal Plane Block Versus Erector Spinae Plane Block in Pediatric Cardiac Patients Undergoing Primary Repair of Septal Defects Via Median Sternotomy
Brief Title: Deep Parasternal Intercostal Plane Block Versus Erector Spinae Plane Block in Pediatric Cardiac Patients Undergoing Primary Repair of Septal Defects Via Median Sternotomy
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sarah Ahmed Hanee Abdelmohaimen Bakr, Assisstant Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMASU MD124/2024
Record Dates: First submitted 2025-02-27; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Septal Defect
Keywords: septal defect; acyanotic heart disease; median sternotomy; deep parasternal intercostal plane block; erector spinae plane block; eras
MeSH Terms: conditions — Heart Septal Defects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Deep Parasternal Intercostal Plane Block (Active Comparator): Patients will receive bilateral deep parasternal intercostal plane block.
  Interventions: Procedure: Deep Parasternal intercostal plane block
- Erector Spinae plane block (Active Comparator): Patients will receive bilateral erector spinae plane block
  Interventions: Procedure: Erector Spinae Plane Block
- conventional analgesic regimen (Active Comparator): patients will receive conventional analgesic regimen
  Interventions: Drug: conventional analgesic regimen

INTERVENTIONS:
Procedure: Deep Parasternal intercostal plane block — Patients will receive bilateral deep parasternal plane block using, 1mg/kg of 0.25% bupivacaine on each side under ultrasound guidance. The total dose of bupivacaine amounting to 2 mg/kg.
  Arms: Deep Parasternal Intercostal Plane Block
Procedure: Erector Spinae Plane Block — Patients will receive bilateral erector spinae plane block using, 1 mg/kg of 0.25% bupivacaine will be administered on each side under ultrasound guidance. The total dose of bupivacaine amounted to 2 mg/kg
  Arms: Erector Spinae plane block
Drug: conventional analgesic regimen — Anesthesia will be induced with IV ketamine, 2 mg/kg, fentanyl, 2 µg/kg, and rocuronium 0.9 mg/kg, administered to facilitate endotracheal intubation.
  Maintenance of anesthesia will be achieved by isoflurane at an end tidal concentration of 1-1.5% in FiO2 of 0.5, intravenous fentanyl at a dose of 1 µg/kg in incremental dosage, and intravenous rocuronium 0.15 mg/kg administration according to nerve stimulator.
  Arms: conventional analgesic regimen

SUMMARY:
In this study we are aiming to compare the Erector Spinae Plane Block and the Deep Parasternal intercostal plane block as regard to their technique, application and outcome in order to describe the most suitable method for pediatric cardiac patients undergoing primary repair of septal defects

The primary outcome of this study will be the time of the first request for postoperative analgesics by FLACC pain scale more than 4 The secondary outcomes will be the total postoperative analgesic consumption, time for extubation, the incidence of nausea and vomiting, hemodynamic instability, onset of ambulation and any other complications on the first day after surgery

Participants will be enrolled in this double-blinded randomly allocated using computer-based randomization into three groups. Group 1 will receive bilateral deep parasternal intercostal plane block. Group 2 will receive bilateral erector spinae plane block. Group 3 will receive conventional analgesic regimen without having a regional block

DETAILED DESCRIPTION:
Pediatric cardiac surgery involving median sternotomy can be associated with significant postoperative pain. Poorly controlled pain following cardiac surgery has been shown to be a risk factor for increased morbidity, including severe cardiopulmonary dysfunction, hypercoagulability, and immunosuppression.

Post-operative pain management, which provides effective analgesia, minimizes side effects and contributes to enhanced recovery after surgery, is a unique challenge in the pediatric cardiac surgery population. The ideal post-operative analgesic regimen would enable early separation from mechanical ventilation, decrease opioid consumption, and expedite discharge from the intensive care unit.

Systemic opioids and non-steroidal anti-inflammatory drugs have been the mainstay for treating pain during the perioperative period in children undergoing median sternotomy for cardiac surgery. The traditional high-dose opioid approach is associated with a decreased stress response but at the expense of prolonged mechanical ventilation, and increased opioid-related side effects. NSAIDs are effective as part of a multimodal analgesic approach, but their use can be limited due to concerns regarding coagulopathy or impairment of renal function.

Regional anesthesia is becoming increasingly popular in pediatric cardiac surgery for its opioid sparing effects. By blocking the afferent impulses from surgical sites, the need for supplemental opioids is reduced. Neuraxial catheters, while effective, are often not utilized in the setting of full heparinization and coagulopathy due to the small yet significant risk of epidural hematoma formation. Paravertebral blocks have similar risk and side effect profiles to neuraxial catheters and require blocks to be performed bilaterally with a posterior approach. Truncal blocks such as erector spinae plane blocks, as well as superficial and deep parasternal blocks, have been shown to provide adequate pain relief for cardiac surgery, and have been gaining popularity.

Appropriate pain relief from a sternotomy incision can be achieved by blocking the second to sixth thoracic intercostal nerves. The newer ultrasound-guided deep parasternal block (previously known as transversus thoracic muscle plane block, involves deposition of a local anesthetic between the internal intercostal and transversus thoracic muscles and effectively blocks the anterior branches of intercostal nerves T2-6.

The recent American Association for Thoracic Surgery Congenital Cardiac Surgery Working Group 2021 consensus document on enhanced recovery after pediatric cardiac surgery gives mention to bilateral transversus thoracic muscle plane blocks (now deep parasternal block) as a regional anesthetic option with opioid-sparing effects but states that more data are needed to determine their efficacy.

On the other hand, Erector spinae plane block is an ultrasound- guided interfascial plane block that has been proposed for the management of thoracic pain. When applied bilaterally, ESPB has been demonstrated to provide effective analgesia at the selected dermatomes including the upper chest (T2-T4) and the mid-chest (T5-T7), which might be useful for postoperative analgesia after cardiac surgery.

In this study, we will compare the use of bilateral single injection deep parasternal blocks versus a second group receiving bilateral single injection erector spinae blocks in pediatric patients undergoing median sternotomy for cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with acyanotic heart disease
* Patients with septal defect undergoing primary repair
* ASA Ⅰ and Ⅱ

Exclusion Criteria:

* Patient's guardian refusal of procedure or participation in the study.
* Patients with hemodynamic instability
* Preexisting infection at the block site
* Allergy to local anesthetics
* Psychiatric illness
* Abnormal coagulation profile
* Preoperative ejection fraction less than 35%
* Recurrent ventricular arrhythmias
* Emergency Surgery
* Redo surgeries

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Time of the first request for postoperative analgesics | 24 hours
  The time of the first request for postoperative analgesics by Face, Legs, Activity, Cry, and Consolability (FLACC) pain scale more than 4.
  Patients will be assessed at 0, ½, 1, 2, 4, 6, 8, 12, 24 hours.

SECONDARY OUTCOMES:
Total postoperative analgesic consumption. | 24 hours
  Comparison between the three groups considering the amount of opioids consumed according to FLACC scale in the post operative period.
Time for extubation | 24 hours
  Comparison between the three groups considering the effect of different pain control modalities on aiding fast track extubation.
Incidence of nausea | 24 hours
  Comparison between the three groups considering the effect of different pain control modalities on the incidence of nausea and vomiting, either by a direct central effect or indirectly due to pain.
Hemodynamic instability | 24 hours
  Comparison between the three groups considering the incidence of hemodynamic instability due to the effect of local anesthetics on hemodynamics or the depressor effect of opioids on the first hours after surgery. Also, the surgical causes of hemodynamic instability in the first day and its effect on the study.
Onset of ambulation | 24 hours
  Comparison between the three groups regarding the onset of ambulation and the effect of the efficacy of pain control in light of early recovery after surgery.
incidence of vomiting | 24 hours
  Comparison between the three groups considering the effect of different pain control modalities on the incidence of nausea and vomiting, either by a direct central effect or indirectly due to pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No